CLINICAL TRIAL: NCT00747084
Title: Can Simple and Inexpensive Techniques Enhance Patient Comfort in Sedation Risk-free Screening and Surveillance Colonoscopy?
Brief Title: Can Simple and Inexpensive Techniques Enhance Patient Comfort
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Instruments necessary to continue project have been removed via medical center staff. Therefore, the project cannot continue until they have been replaced.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: FLVA0055
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Colonoscopy
Keywords: unsedated colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Study Treatment (Experimental): Study Treatment: warm water loading of the sigmoid colon and warm water irrigation for dealing with colonic spasms.
  Interventions: Procedure: Colonoscopy
- Arm 2: Control Treatment (No Intervention): Control Treatment: no water loading and waiting for spasms to subside.

INTERVENTIONS:
Procedure: Colonoscopy — The purpose of the study is to conduct an RCT study to determine the effectiveness of loading the sigmoid colon with warm water and warm water irrigation for dealing with colonic spasms in enhancing patient abdominal comfort during unsedated colonoscopy.
  Arms: Arm 1: Study Treatment

SUMMARY:
This research study compares two methods of performing colonoscopy without sedation. The standard method is to insert the colonoscope without adding any water to the colon, and when colonic spasms occur during the examination, waiting for the spasms to subside before continuing with the insertion of the colonoscope. The study method involves putting 200 ml (7 oz) of warm water through the colonoscope into the colon at the beginning of the examination, and when colonic spasms occur during the examination, putting 30 ml (1 oz) of warm water into the spastic area(s) to relax the colonic spasms.

DETAILED DESCRIPTION:
The purpose of the study is to conduct a RCT study to determine the effectiveness of loading the sigmoid colon with warm water and warm water irrigation for dealing with colonic spasms in enhancing patient abdominal comfort during unsedated colonoscopy. The specific aim is to compare Study Treatment of warm water loading and irrigation when spasms occur with Control Treatment of no water loading and waiting for spasms to subside. The proportion of patients complaining of abdominal discomfort and their discomfort score are the primary outcome variables. The secondary outcome variables and co-variables described below will be recorded in a prospective manner to ensure completeness of data collection. In preliminary clinical observation at VA Sepulveda ACC, 25 to 30% of VA patients accept colonoscopy without sedation. The goal of this study is to find ways of further reducing discomfort associated with unsedated colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female
* Adult patients 18 years old in need of colonoscopy for screening or follow up of colonic polyps, and willing to consent to be randomized.

Exclusion Criteria:

* Patients receiving outpatient prescription narcotic treatment [more likely to have discomfort response even with sedation (42)].
* Patients who report excessive anxiety [pre-endoscopy appointment, single question asking how anxious the patient generally is, four point scale (1 = not at all, 2 = slightly, 3 = moderately, 4 = excessively].
* Excessive anxiety is significantly correlated with lack of cooperation during colonoscopy and high dissatisfaction score after the procedure (43).
* Patients with moderate to severe abdominal discomfort, unable to provide informed consent, have a poor bowel preparation (discolored rectal output or feces filled rectal vault), and those who decline to participate, will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare Study Treatment of warm water loading and irrigation when spasms occur with Control Treatment of no water loading and waiting for spasms to subside. The proportion of patients complaining of abdominal discomfort and their discomfort score are | Immediately after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Felix W Leung, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- [Derived] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405